CLINICAL TRIAL: NCT04674189
Title: COVID-19: A Phase 3, Randomized, Observer-Blinded, Placebo-Controlled Clinical Study Evaluating the Safety and Immunogenicity of Investigational SARS-CoV-2 mRNA Vaccine CVnCoV in Adult Health Care Workers in Mainz (Germany)
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Vaccine CVnCoV in Healthy Adults in Germany for COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CureVac (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV-NCOV-005
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2022-02

CONDITIONS: Coronavirus; Covid19; SARS-CoV-2; Severe Acute Respiratory Syndrome
Keywords: Vaccine; SARS; COVID; Safety; Immunogenicity
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Severe Acute Respiratory Syndrome | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CVnCoV: Group 1, Lot 1 (Experimental): Participants in Group 1 will be vaccinated with CVnCoV 12 µg mRNA on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV Vaccine
- CVnCoV: Group 2, Lot 2 (Experimental): Participants in Group 2 will be vaccinated with CVnCoV 12 µg mRNA on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Biological: CVnCoV Vaccine
- Placebo (Placebo Comparator): Participants will receive a placebo on Day 1 and Day 29 in the deltoid area, preferably in the non-dominant arm.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CVnCoV Vaccine — Intramuscular injection
  Other Names: CV07050101
  Arms: CVnCoV: Group 1, Lot 1; CVnCoV: Group 2, Lot 2
Drug: Placebo — Intramuscular injection
  Arms: Placebo

SUMMARY:
This study aims to evaluate the safety (in all participants) and reactogenicity (in a subset of participants) of CVnCoV administered as a 2-dose schedule to adult participants 18 years of age or older. The study also aims to assess antibody responses to the receptor-binding domain (RBD) of spike (S) protein of SARS-CoV-2 after 1 and 2 doses of CVnCoV in adults 18 years of age or older included in a subset of participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants 18 years of age or older.
* Health care workers (HCWs), employees or students in clinical training.
* Provide written informed consent prior to initiation of any trial procedures.
* Expected compliance with protocol procedures and availability for clinical follow-up through the last planned visit.
* Females of non-childbearing potential defined as follows: surgically sterile (history of bilateral tubal ligation/occlusion, bilateral oophorectomy or hysterectomy) or postmenopausal (defined as amenorrhea for ≥12 consecutive months prior to screening [Day 1] without an alternative medical cause). A follicle-stimulating hormone (FSH) level may be measured at the discretion of the investigator to confirm postmenopausal status.
* Females of childbearing potential: negative urine pregnancy test (human chorionic gonadotropin within 24 hours prior to each trial vaccination on Day 1 and Day 29.
* Females of childbearing potential must use highly effective methods of birth control from 2 weeks before the first administration of the trial vaccine until 3 months following the last administration. The following methods of birth control are considered highly effective when used consistently and correctly:

  * Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal or transdermal);
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable or implantable);
  * Intrauterine devices (IUDs);
  * Intrauterine hormone-releasing systems (IUSs);
  * Bilateral tubal ligation;
  * Vasectomized partner;
  * Sexual abstinence (periodic abstinence [e.g., calendar, ovulation, symptothermal and post-ovulation methods] and withdrawal are not acceptable).

Exclusion Criteria:

* History of virologically confirmed SARS-CoV-2 infection or SARS-CoV-2 positive serology.
* For females: pregnancy or lactation.
* Use of any investigational or non-registered product (vaccine or drug) within 28 days preceding the administration of the first trial vaccine or planned use during the trial.
* Receipt of licensed vaccines within 28 days (for live vaccines) or 14 days (for inactivated vaccines) prior to the administration of trial vaccine.
* Prior administration of any investigational SARS-CoV-2 vaccine or other coronavirus (SARS-CoV, MERS-CoV) vaccine or planned use during the trial.
* Any treatment with immunosuppressants or other immune-modifying drugs (including but not limited to corticosteroids, biologicals and methotrexate) for > 14 days total within 6 months preceding the administration of trial vaccine or planned use during the trial. For corticosteroid use, this means prednisone or equivalent, 0.5 mg/kg/day for 14 days or more. The use of inhaled, topical, or localized injections of corticosteroids (e.g., for joint pain/inflammation) is permitted.
* Any medically diagnosed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination including known infection with human immunodeficiency virus (HIV), current diagnosis of or treatment for cancer including leukemia, lymphoma, Hodgkin disease, multiple myeloma or generalized malignancy; chronic renal failure or nephrotic syndrome; and receipt of an organ or bone marrow transplant.
* Active or chronic disease of, or currently on treatment for, hepatitis B virus (HBV) or hepatitis C virus (HCV).
* History of angioedema (hereditary or idiopathic), or a history of any anaphylactic reaction.
* History of Potential immune-mediated disease (pIMD).
* History of allergy to any component of CVnCoV vaccine.
* Administration of immunoglobulins or any blood products within 3 months prior to the administration of trial vaccine, or planned receipt during the trial.
* Participants with a significant acute or chronic medical or psychiatric illness that, in the opinion of the investigator, precludes trial participation (e.g., may increase the risk of trial participation, render the participant unable to meet the requirements of the trial, or may interfere with the participant's trial evaluations). These include severe and/or un-controlled cardiovascular disease, gastrointestinal disease, liver disease, renal disease, respiratory disease, endocrine disorder, and neurological and psychiatric illnesses.
* Participants with impaired coagulation or any bleeding disorder in whom an intramuscular (IM) injection or a blood draw is contraindicated. However, those with controlled and stable cases can be included in the trial.
* Foreseeable non-compliance with protocol as judged by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2357 (Actual)
Dates: Start 2020-12-23 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsmedizin der Johannes-Gutenberg-Universität Mainz Langenbeckstr. 1, Mainz, Germany

REFERENCES:
- [Derived] Kowalzik F, Teschner D, Mesquita M, Jensen C, Schreiner D, Kronfeld K, Tubic-Grozdanis M, Cheatham-Seitz D, Hettich F, Quintini G, Schoenborn-Kellenberger O, Codo P, von Eisenhart-Rothe P, Mann P, Oostvogels L, Gehring S. A phase 3, randomised, observer-blinded, placebo controlled-trial evaluating the safety and immunogenicity of investigational SARS-CoV-2 mRNA vaccine CVnCoV in adult healthcare workers in Mainz (Germany). Vaccine X. 2024 Jun 20;19:100512. doi: 10.1016/j.jvacx.2024.100512. eCollection 2024 Aug. PMID 39040887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was performed in Germany between 23 December 2020 and 08 June 2022.
Pre-assignment Details: Of the 2357 participants who were randomized, 2351 participants were treated.
Groups:
- CVnCoV: Group 1, Lot 1: Participants in Group 1 were vaccinated with CVnCoV 12 µg Lot 1 as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
- CVnCoV: Group 2, Lot 2: Participants in Group 2 were vaccinated with CVnCoV 12 µg Lot 2 as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
- Placebo: Participants received a placebo as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
Period: Overall Study
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Started | 786 | 786 | 785
Safety Analysis Set | 783 | 785 | 783
Completed | 617 | 637 | 372
Not Completed | 169 | 149 | 413
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Received Alternative Authorized Vaccine | 0 | 1 | 17
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Withdrawal by Participant | 83 | 71 | 142
Not completed — Lost to Follow-up | 55 | 53 | 44
Not completed — Miscellaneous | 27 | 23 | 207
Not completed — Did Not Receive Treatment | 3 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants randomized in the trial who received at least one dose of any lot of CVnCoV or placebo vaccine.
Groups:
- Total: Total of all reporting groups
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo | Total
Number analyzed (Participants) | 783 | 785 | 783 | 2351
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.2 (14.88) | 43.4 (14.80) | 42.7 (14.52) | 42.7 (14.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 527 | 539 | 521 | 1587
  Male | 256 | 246 | 262 | 764
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 4 | 14
  Not Hispanic or Latino | 764 | 759 | 758 | 2281
  Unknown or Not Reported | 14 | 21 | 21 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 755 | 765 | 760 | 2280
  Black or African American | 2 | 1 | 0 | 3
  Asian | 13 | 9 | 14 | 36
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Other | 4 | 3 | 5 | 12
  Unknown or Not Reported | 7 | 6 | 4 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Medically Attended Adverse Event (AE) Occurring in the Following 6 Months After Dose 2
Description: Medically attended AEs were defined as AEs with medically attended visits that are not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AE.
Time Frame: Up to 6 months after Dose 2 (Days 29 to 211)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants
  Any medically attended AEs | 95 | 133 | 58
  Any related medically attended AEs | 34 | 32 | 13

2. Primary Outcome: Number of Participants Who Experienced a Serious Adverse Event (SAE)
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AE.
Time Frame: Day 1 to Day 393
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants
  Any SAEs | 8 | 10 | 6
  Any related SAEs | 1 | 1 | 0

3. Primary Outcome: Intensity of SAEs Per the Investigator's Assessment
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
  The Investigator made an assessment of intensity for each AE reported during the trial and assigned it to one of the following categories:
  * Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  * Moderate: an event that caused sufficient discomfort to interfere with normal everyday activities.
  * Severe: an event that prevented normal everyday activities.
Time Frame: Day 1 to Day 393
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants
  Any mild SAEs | 0 | 0 | 0
  Any moderate SAEs | 2 | 5 | 1
  Any severe SAEs | 6 | 5 | 5

4. Primary Outcome: Number of Participants Who Experienced an Adverse Event of Special Interest (AESI) Occurring in the Following 1 Year After Dose 2
Description: The following events were considered and collected as AESI throughout the trial:
  * AEs with a suspected immune-mediated etiology.
  * Other AEs relevant to SARS-CoV-2 vaccine development or the target disease.
  * COVID-19.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AE.
Time Frame: Up to 1 year after Dose 2 (Days 29 to 393)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants
  Any AESIs | 14 | 14 | 5
  Any related AESIs | 7 | 5 | 0

5. Primary Outcome: Number of Participants Who Experienced Death Due to SAE
Description: An SAE was defined as any untoward medical occurrence that, at any dose:
  * Resulted in death.
  * Was life-threatening.
  * Required inpatient hospitalization or prolongation of existing hospitalization.
  * Resulted in persistent disability/incapacity.
  * Was a congenital anomaly/birth defect in the offspring of the participant.
  * Was an important medical event.
Time Frame: Day 1 to Day 393
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants | 0 | 0 | 0

6. Primary Outcome: Number of Participants Who Experienced an AE Leading to Vaccine Withdrawal Occurring in the Following 1 Year After Dose 2
Time Frame: Up to 1 year after Dose 2 (Days 29 to 393)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants | 7 | 5 | 2

7. Primary Outcome: Number of Participants Who Experienced an AE Leading to Trial Discontinuation Occurring in the Following 1 Year After Dose 2
Time Frame: Up to 1 year after Dose 2 (Days 29 to 393)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 783 | 785 | 783
Participants | 1 | 0 | 1

8. Primary Outcome: Number of Participants Who Experienced an Unsolicited AE Occurring on the Day of Vaccination and the Following 28 Days After Any Dose
Description: eDiaries were used for the collection of unsolicited AEs on each vaccination day and the following 28 days.
  The Investigator assessed the relationship between trial vaccine and occurrence of each AE.
Time Frame: Day 1 to 28 days after Dose 2 (Day 57)
Population: Safety Analysis Subset: The first 1289 participants enrolled who belong to the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 430 | 429 | 430
Participants
  Any unsolicited AEs | 245 | 270 | 187
  Any related unsolicited AEs | 183 | 186 | 88

9. Primary Outcome: Intensity of Unsolicited AEs Per the Investigator's Assessment Occurring on the Day of Vaccination and the Following 28 Days After Any Dose
Description: eDiaries were used for the collection of unsolicited AEs on each vaccination day and the following 28 days.
  The Investigator made an assessment of intensity for each AE reported during the trial and assigned it to one of the following categories:
  * Mild: an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
  * Moderate: an event that caused sufficient discomfort to interfere with normal everyday activities.
  * Severe: an event that prevented normal everyday activities.
Time Frame: Day 1 to 28 days after Dose 2 (Day 57)
Population: Safety Analysis Subset: The first 1289 participants enrolled who belong to the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
Number analyzed (Participants) | 430 | 429 | 430
Participants
  Any mild unsolicited AEs | 133 | 149 | 114
  Any moderate unsolicited AEs | 73 | 71 | 42
  Any severe unsolicited AEs | 14 | 28 | 10
  Any unsolicited AEs without intensity assessment | 25 | 22 | 21

10. Primary Outcome: Occurrence of Seroconversion for SARS-CoV-2 Receptor-Binding Domain (RBD) of Spike Protein Antibodies (IgG) on Day 29 and Day 43
Description: Titers of IgG antibodies directed against the SARS-CoV-2 RBD of Spike Protein antigen were measured by enzyme-linked immunosorbent assay (ELISA). Percentage with 95% confidence interval (CI) of participants for whom a seroconversion was observed is presented by group. Seroconversion was defined as a fold increase above 1 in SARS-CoV-2 Spike Protein RBD IgG antibody levels in participants seronegative at Baseline. Participants who tested positive for COVID-19 had their data included up to the point of a positive test result. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline (Day 1), Day 29 and Day 43
Population: Per Protocol Immunogenicity Set: 250 participants who received both doses as randomized and within the windows defined in the protocol, had no major protocol deviations expected to impact the immunogenicity outcomes, and had not received medical treatments that may interfere with any of the immunogenicity measurements. Only participants seronegative at Baseline with evaluable samples at each visit are included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CVnCoV: Pooled Lots 1 and 2: Participants in Group 1 and Group 2. Participants were vaccinated with either CVnCoV 12 µg Lot 1 or CVnCoV 12 µg Lot 2 as an intramuscular injection by needle in the deltoid area on Day 1 and Day 29.
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | CVnCoV: Pooled Lots 1 and 2 | Placebo
Number analyzed (Participants) | 99 | 98 | 197 | 48
percentage of participants
  Day 29 | 8.1 [3.6 to 15.3] | 18.4 [11.3 to 27.5] | 13.2 [8.8 to 18.7] | 0.0 [0.0 to 7.4]
  Day 43: number analyzed (Participants) | 88 | 86 | 174 | 41
  Day 43 | 95.5 [88.8 to 98.7] | 94.2 [87.0 to 98.1] | 94.8 [90.4 to 97.6] | 0.0 [0.0 to 8.6]

11. Primary Outcome: SARS-CoV-2 RBD of Spike Protein Antibody (IgG) Levels on Days 1, 29 and 43
Description: Titers of IgG antibodies directed against the SARS-CoV-2 RBD of Spike Protein antigen were measured by ELISA and expressed as geometric mean of titers (GMT) with 95% CI, by group. Individual values below the lower limit of quantification (LLOQ) were set to half of the LLOQ. Participants who tested positive for COVID-19 had their data included up to the point of a positive test result. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 1, Day 29 and Day 43
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | CVnCoV: Pooled Lots 1 and 2 | Placebo
Number analyzed (Participants) | 99 | 98 | 197 | 48
GMT
  Day 1 | 50.000 [50.000 to 50.000] | 50.000 [50.000 to 50.000] | 50.000 [50.000 to 50.000] | 50.000 [50.000 to 50.000]
  Day 29 | 55.145 [51.403 to 59.160] | 62.236 [56.437 to 68.631] | 58.566 [55.144 to 62.199] | 50.000 [50.000 to 50.000]
  Day 43: number analyzed (Participants) | 88 | 86 | 174 | 41
  Day 43 | 1285.722 [1003.885 to 1646.683] | 1151.416 [869.345 to 1525.008] | 1217.489 [1011.594 to 1465.289] | 50.000 [50.000 to 50.000]

12. Secondary Outcome: Occurrence of Seroconversion for SARS-CoV-2 Neutralizing Antibodies on Day 29 and Day 43
Description: Neutralizing activity of induced antibodies was determined by an activity assay. Percentage with 95% CI of participants for whom a seroconversion was observed is presented by group. Seroconversion was defined as a fold increase above 1 in SARS-CoV-2 neutralizing antibody levels in participants seronegative at Baseline. Participants who tested positive for COVID-19 had their data included up to the point of a positive test result. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Baseline (Day 1), Day 29 and Day 43
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | CVnCoV: Pooled Lots 1 and 2 | Placebo
Number analyzed (Participants) | 99 | 98 | 197 | 48
percentage of participants
  Day 29 | 2.0 [0.2 to 7.1] | 2.0 [0.2 to 7.2] | 2.0 [0.6 to 5.1] | 0.0 [0.0 to 7.4]
  Day 43: number analyzed (Participants) | 88 | 86 | 174 | 41
  Day 43 | 76.1 [65.9 to 84.6] | 75.6 [65.1 to 84.2] | 75.9 [68.8 to 82.0] | 0.0 [0.0 to 8.6]

13. Secondary Outcome: SARS-CoV-2 Neutralizing Antibody Levels on Days 1, 29 and 43
Description: Neutralizing activity of induced antibodies was determined by an activity assay. GMT with 95% CI of SARS-CoV-2 neutralizing antibody levels is presented by group. Individual values below the LLOQ were set to half of the LLOQ. Participants who tested positive for COVID-19 had their data included up to the point of a positive test result. Participants who received a licensed/authorized vaccine were censored at the day after receiving the licensed/authorized vaccine.
Time Frame: Day 1, Day 29 and Day 43
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | CVnCoV: Pooled Lots 1 and 2 | Placebo
Number analyzed (Participants) | 99 | 98 | 197 | 48
GMT
  Day 1 | 5.000 [5.000 to 5.000] | 5.000 [5.000 to 5.000] | 5.000 [5.000 to 5.000] | 5.000 [5.000 to 5.000]
  Day 29 | 5.160 [4.906 to 5.427] | 5.071 [4.972 to 5.172] | 5.116 [4.980 to 5.256] | 5.000 [5.000 to 5.000]
  Day 43: number analyzed (Participants) | 88 | 86 | 174 | 41
  Day 43 | 28.846 [21.716 to 38.318] | 23.976 [18.394 to 31.252] | 26.327 [21.707 to 31.929] | 5.000 [5.000 to 5.000]

ADVERSE EVENTS:
Time Frame: Day 1 to Day 393
Description: Safety Analysis Set: All participants randomized in the trial who received at least one dose of any lot of CVnCoV or placebo vaccine.
Arm/Group | CVnCoV: Group 1, Lot 1 | CVnCoV: Group 2, Lot 2 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/783 | 0/785 | 1/783
Serious Adverse Events (participants affected / at risk) | 8/783 | 10/785 | 6/783
Other Adverse Events (participants affected / at risk) | 542/783 | 547/785 | 475/783
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVnCoV: Group 1, Lot 1 (N=783) | CVnCoV: Group 2, Lot 2 (N=785) | Placebo (N=783)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Small intestine gangrene (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0)
Ganglioglioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CVnCoV: Group 1, Lot 1 (N=783) | CVnCoV: Group 2, Lot 2 (N=785) | Placebo (N=783)
Diarrhoea (Gastrointestinal disorders) | 104 (146) | 113 (144) | 66 (78)
Nausea (Gastrointestinal disorders) | 140 (197) | 132 (195) | 65 (82)
Chills (General disorders) | 276 (419) | 275 (457) | 81 (95)
Fatigue (General disorders) | 425 (835) | 427 (852) | 278 (530)
Injection site pain (General disorders) | 387 (693) | 390 (698) | 160 (205)
Injection site pruritus (General disorders) | 27 (31) | 43 (53) | 18 (22)
Pyrexia (General disorders) | 218 (309) | 221 (330) | 61 (64)
Arthralgia (Musculoskeletal and connective tissue disorders) | 250 (376) | 245 (378) | 75 (98)
Myalgia (Musculoskeletal and connective tissue disorders) | 344 (569) | 341 (565) | 136 (183)
Dizziness (Nervous system disorders) | 37 (42) | 46 (54) | 34 (43)
Headache (Nervous system disorders) | 428 (924) | 430 (952) | 293 (615)
Cough (Respiratory, thoracic and mediastinal disorders) | 70 (89) | 85 (106) | 62 (84)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 98 (128) | 106 (145) | 95 (121)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 106 (134) | 107 (135) | 99 (133)
Pain (General disorders) | 46 (53) | 62 (68) | 47 (52)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 32 (38) | 39 (44) | 41 (47)
COVID-19 (Infections and infestations) | 106 (111) | 99 (103) | 123 (131)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/89/NCT04674189/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/89/NCT04674189/SAP_001.pdf